CLINICAL TRIAL: NCT03499392
Title: Primary Headache and Psychological Factors, Mental Functioning and Attachment Modalities.
Acronym: CEPRIVA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: P/2017/344
Record Dates: First submitted 2018-01-16; First posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-03

CONDITIONS: Primary Headache Disorder
Keywords: psychological factors
MeSH Terms: conditions — Headache Disorders, Primary | interventions — Psychological Tests; Interview, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- psychological investigation (Other)
  Interventions: Other: psychological tests

INTERVENTIONS:
Other: psychological tests — psychological tests psychological interviews
  Other Names: psychological interviews

SUMMARY:
The World Health Organization (WHO) ranks headache among the top 20 causes of disability in the world.

Primary headaches (with no known organic cause) account for 90% of these conditions. INSERM estimates that 15% of the general population is concerned. WHO estimates that 1.7-4% of the global adult population is affected by headache for at least 15 days a month. Headaches are disabling, for patients (pain, suffering, fatigue, unavailability ...) but also for society (socio-economic cost as frequent work stoppages and drug costs). They are a public health problem.

In 2002, the High Authority of Health published its recommendations for the diagnosis and management of migraine patients. In addition, the French Society for Migraine and Headache Studies updated these recommendations in 2013. They are focused on the medical management offered by doctors and pharmacists. However, the professionals in daily contact with the subjects know that the dimension psychic plays an important role in the etiology of headaches.

DETAILED DESCRIPTION:
The review of the literature shows the keen interest and the need for this type of research to better understand the main psychological factors involved in primary headaches.

The current vagueness, the lack of knowledge regarding the aspects associated psychological and the lack of studies on the French population can be filled with this study which takes place at the University Hospital of Besançon.

ELIGIBILITY:
Inclusion Criteria:

* first consultation in neurology good general somatic state

Exclusion Criteria:

* Pregnancy History of psychiatric disorder

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-04-30 (Actual); Primary Completion 2018-04-30 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of headache attacks | Month 9
  Symptomatic evolution assessed with a composite outcome (number of episodes + severity of headaches) reported by patient and collected during neurological consultation
Duration of each headache attack | Month 9
  Symptomatic evolution assessed with a composite outcome (number of episodes + duration of each episode) reported by patient and collected during neurological consultation

SECONDARY OUTCOMES:
Definition of patient's psychological profile | Month 9
  Profile is determined by additional semi-structured interviews + Rorschach test + Adult Attachment Interview + mini-Social cognition and Emotional Assesment test (qualitative outcomes).

CONTACTS AND LOCATIONS:
Locations (1):
- Belot, Besançon, Doubs, France